CLINICAL TRIAL: NCT06557057
Title: Impact of Aromatase Inhibitor Therapy on Glucose Homeostasis and Diabetes Risk
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-005595; NCI-2024-01190 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-005595 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: HER2-Positive Breast Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples retained for future research with permission of participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood sample collection, glucose testing, DEXA scan to measure body composition, complete a questionnaire and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
This study assesses the effect of hormone directed treatment for breast cancer on glucose metabolism.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the impact of endocrine adjuvant therapy with aromatase inhibitors in women with hormone receptor positive breast cancer or ductal carcinoma in situ (DCIS) on various indices of glucose homeostasis, utilizing oral minimal model assessment, in comparison to healthy post menopausal women and another cohort of women on tamoxifen.

OUTLINE: This is an observational study.

Patients undergo blood sample collection, glucose testing, dual-energy x-ray absorptiometry (DEXA)scan to measure body composition, complete a questionnaire and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women with hormone receptor positive breast cancer or ductal carcinoma in situ (DCIS). Post-menopause will be defined as women who experience 12 months of amenorrhea or have undergone bilateral salpingo-oophorectomy.

  * 25 women who are planning to start or are within 6 months of starting treatment with aromatase inhibitors, after consultation in breast clinic and cancer center.
  * 25 women who will be starting Tamoxifen (comparative group)
  * 25 healthy post menopausal women will also be recruited.

Exclusion Criteria:

* Established diagnosis of diabetes
* Therapy with medications that could affect glucose metabolism
* Screening fasting glucose ≥ 126 mg/dl, and/or HbA1c ≥ 6.5%
* History of upper GI surgery that alters gastric emptying or causing malabsorption e.g., bariatric surgery, fundoplication

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Post-menopausal women with hormone receptor positive breast cancer or DCIS who are planning to start or within 6 months of starting treatment with an aromatase inhibitor or tamoxifen and healthy post-menopausal women.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Disposition Index (DI) | Baseline; up to 1 year
  Will be calculated as the product of beta cell responsivity and Si (insulin action). DI of women with hormone receptor positive breast cancer or DCIS treated with aromatase inhibitors will be compared to DI of healthy post menopausal women. Participants will undergo a history, physical examination, and a blood collection for fasting glucose, and Hemoglobin A1C (HbA1c) at baseline and one year later. Participants will be contacted at 3 and 6 months by phone to confirm continued use of the endocrine therapy that was initiated by the clinical team.
Glucose homeostasis - tamoxifen compared to no treatment | Baseline; up to 1 year
  Glucose homeostasis is the process by which the body regulates blood glucose levels, also known as blood sugar, within a narrow range. Glucose homeostasis of women with hormone receptor positive breast cancer or DCIS treated with tamoxifen will be compared to glucose homeostasis of women without treatment. Participants will undergo a history, physical examination, and a blood collection for fasting glucose, and Hemoglobin A1C (HbA1c) at baseline and one year later. Participants will be contacted at 3 and 6 months by phone to confirm continued use of the endocrine therapy that was initiated by the clinical team.
Glucose homeostasis - aromatase inhibitor compared to tamoxifen | Baseline; up to 1 year
  Glucose homeostasis is the process by which the body regulates blood glucose levels, also known as blood sugar, within a narrow range. Glucose homeostasis of women with hormone receptor positive breast cancer or DCIS treated with aromatase inhibitors will be compared to glucose homeostasis of women treated with tamoxifen. Participants will undergo a history, physical examination, and a blood collection for fasting glucose, and Hemoglobin A1C (HbA1c) at baseline and one year later. Participants will be contacted at 3 and 6 months by phone to confirm continued use of the endocrine therapy that was initiated by the clinical team.

CONTACTS AND LOCATIONS:
Overall Officials: Kalpana Muthusamy, MBBS, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials